CLINICAL TRIAL: NCT00710177
Title: Prostaglandin G/H Synthase-1 (PTGS1) Genetic Variation and Increased Risk for Persistent Pulmonary Hypertension of the Newborn (PPHN)
Brief Title: PTGS1 Genetic Variation and Increased Risk for Persistent Pulmonary Hypertension of the Newborn
Acronym: PPHN
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, G. Ganesh Konduri, Chair, Division of Neonatology, Medical College of Wisconsin
Other Study IDs: PRO46055
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
Keywords: PPHN; PTGS1; NSAID
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, meconium
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PPHN: Infants born at >= 34 weeks who are diagnosed with clinical and/or echocardiographic evidence of PPHN
- Control: Randomly selected, normal healthy infants born at >= 34 weeks gestational age and do not have PPHN

SUMMARY:
The purpose of this study is to determine if normally occurring variations in a specific gene called PTGS-1 are associated with an increased risk of narrowing of the ductus arteriosus from exposure to over-the-counter pain medicines (NSAIDs).

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of the newborn (PPHN) occurs when the pulmonary vascular resistance fails to decrease at birth during the transition to postnatal life. The affected infants have severe hypoxemia, a 10% risk of mortality, and among survivors, a 30% incidence of long term neurodevelopmental and hearing deficits. The etiology of PPHN in the majority of affected infants remains unknown. Although constriction of fetal ductus arteriosus in response to maternal intake of non-steroidal anti-inflammatory drugs (NSAID) has been implicated in PPHN case reports, our laboratory was the first to provide objective evidence for such an association. Nearly 87% of infants with PPHN were exposed to NSAID in utero. Yet 25% of control infants also were exposed without developing PPHN. The basis for the biological susceptibility of some neonates to in utero NSAID exposure remains poorly understood. The hypothesis of this proposal is that PTGS1 genetic variation is associated with increased susceptibility to ductal constriction from in utero NSAID exposure and an increased risk of PPHN. This hypothesis will be tested through the following specific aims: Determine the incidence of PTGS1 sequence variants in PPHN patients versus matched controls. PTGS1 sequence will include all 11 exons, a minimum of 100 bp of exon flanking sequences, and 1 kbp of upstream regulatory information. Cycle sequencing will be performed followed by analysis using capillary electrophoresis. Differences in the frequency of sequence variants will be determined using Fisher's exact test. The study will also quantify NSAID exposure in meconium samples using a previously established GC/MS assay and correlate exposure levels to both the incidence of PPHN and the presence or absence of PTGS1 sequence variants using regression analysis. Benefits include the ability to predict risk for PPHN based on PTGS1 sequence and avoidance of such risk in the future, thereby reducing patient morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Infants born greater than or equal to 34 weeks gestational age diagnosed with PPHN and normal, healthy infants born greater than or equal to 34 weeks gestational age.

Exclusion Criteria:

* Patients will be excluded if they are diagnosed with lethal congenital anomalies
* structural congenital heart disease except presence of patent ductus arteriosus (PDA) or patent foramen ovale
* structural gastrointestinal tract abnormality that could interfere with meconium passage
* congenital anomalies such as diaphragmatic hernia, Potter's syndrome, or pulmonary hypoplasia

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants born greater than or equal to 34 weeks gestational age diagnosed with PPHN and normal, healthy infants born greater than or equal to 34 weeks gestational age.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether or not a variation in the prostaglandin G/H Synthase-1 gene contributes to the incidence of PPHN in infants who are exposed to NSAIDs in utero. | participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: G. Ganesh Konduri, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No